CLINICAL TRIAL: NCT01762072
Title: Effect of Vitamin B12 and n-3 Polyunsaturated Fatty Acids on Plasma Homocysteine
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, Tao Huang, postdoctoral researcher, Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: No.30972464
Record Dates: First submitted 2013-01-02; First posted 2013-01-07 (Estimated); Last update posted 2013-01-07 (Estimated); Status verified 2013-01

CONDITIONS: Healthy
Keywords: homocysteine-vitamin B12-fish oil-ferritin
MeSH Terms: interventions — Fish Oils

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- vitaminB12 (Placebo Comparator): VitB12 group (VitB12, n=10) receives 8 weeks of treatment with daily oral doses of 1000 μg of vitamin B12 (one capsule)
  Interventions: Dietary Supplement: vitaminB12
- Fish oil (Experimental): Fish oil group (FO, n=10)receives 8 weeks of treatment with daily oral doses of 2g of fish oil in the form of two capsules of fish oil) .
  Interventions: Dietary Supplement: Fish oil
- Fish oil+vitaminB12 (Experimental): VitB12+Fish oil group (VitB12+FO, n=10) receives 8 weeks of treatment with daily oral doses of a combination of 1000 μg of vitamin B12 and 2g of fish oil
  Interventions: Dietary Supplement: Fish oil; Dietary Supplement: vitaminB12

INTERVENTIONS:
Dietary Supplement: Fish oil
  Arms: Fish oil; Fish oil+vitaminB12
Dietary Supplement: vitaminB12
  Arms: Fish oil+vitaminB12; vitaminB12

SUMMARY:
Vitamin B12and n-3 polyunsaturated fatty acids (PUFA) decrease blood homocysteine (Hcy) concentration. However, the combined effect of these nutrients on Hcy and ferritin, and C-reactive protein is limited and inconclusive. The objective was to examine the synergistic effect of vitamin B12 in combination of n-3 PUFA on plasma Hcy, ferritin, and other biochemical markers. In a randomized controlled trial, thirty eligible subjects were randomly divided into three groups, and assigned to receive 1000 μg of vitamin B12, 2g fish oil, or 1000 μg vitamin B12 and 2g fish oil respectively for 8 weeks. Plasma phospholipid (PL) fatty acids and biochemical markers were determined. we hypothesize that combination of vitamin B12 and fish oil have synergistic effect on lowering plasma concentrations of Hcy and ferritin.

ELIGIBILITY:
Inclusion Criteria:

* reliability, regular eating habits, normal weight, nondrinking, and nonsmoking status

Exclusion Criteria:

* None of the selected subjects used any vitamins or dietary supplements and was taking no medication for at least 8 weeks before the start of and during the entire experimental period

Ages: 20 Years to 28 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2013-01; Primary Completion 2013-03 (Estimated)

PRIMARY OUTCOMES:
homocysteine,umol/L | 10 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Zhejiang university, Hangzhou, Zhejiang, China

REFERENCES:
- [Derived] Huang T, Li K, Asimi S, Chen Q, Li D. Effect of vitamin B-12 and n-3 polyunsaturated fatty acids on plasma homocysteine, ferritin, C-reaction protein, and other cardiovascular risk factors: a randomized controlled trial. Asia Pac J Clin Nutr. 2015;24(3):403-11. doi: 10.6133/apjcn.2015.24.3.19. PMID 26420180